CLINICAL TRIAL: NCT04666428
Title: An Observational Study to Determine the Effects of Human Papillomavirus Diagnosis on Relationships of Head and Neck Cancer Patients
Brief Title: Effects of Human Papillomavirus Diagnosis on Relationships of Patients With Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 19D.927; JT 14649 (Other: JeffTrial Number)
Record Dates: First submitted 2020-03-16; First posted 2020-12-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial studies the effects of human papillomavirus diagnosis on the relationships of patients with head and neck cancer. Determining the effects of human papillomavirus diagnosis on relationships may determine whether human papillomavirus-positive patients and their partners are more likely to experience decline in relationship intimacy after diagnosis than human papillomavirus-negative patients and their partners. This may help researchers provide valuable insight into the degree to which a diagnosis of human papillomavirus affects patient relationships over and above the effects of a cancer diagnosis and address the need for additional patient counseling or education following diagnosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the agreement between patients' perceived intimacy level and their partners' perceived intimacy level at different time points in the course of their head and neck cancer (HNC) treatment.

II. To compare any changes in the patients' perceived intimacy scores between human papillomavirus (HPV)-positive and HPV-negative HNC patients at different time points in the course of their HNC treatment.

EXPLORATORY OBJECTIVE:

I. Identify areas of concern or misinformation among patients and partners where further patient counseling or education may be indicated.

OUTLINE:

Patients and partners complete surveys over 10 minutes prior to surgery and 3-6 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Diagnosis of head and neck cancer (previously untreated, any stage) or in a partnered relationship with an individual diagnosed with head and neck cancer
* Tumors positive for HPV
* Tumors negative for HPV
* Treatment plan is intent to cure
* In a partnered relationship
* Willing to answer brief survey prior to treatment and again after completion of treatment
* English Speaking

Exclusion Criteria:

* Prior treatment (surgery, chemotherapy, radiation therapy [XRT], or chemoradiotherapy [CRT]) for head and neck cancer
* Partners of eligible patients undergoing active cancer treatment
* Not in a partnered relationship
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HNC and their partners at Thomas Jefferson University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Change in patients' and partners' perceived intimacy scores at baseline | Before treatment
  Defined as total scores of the primary questions in patient survey and partner survey
Change in patients' and partners' perceived intimacy scores post treatment | within 30 weeks after treatment
  Defined as total scores of the primary questions in patient survey and partner survey
Change Patients' and partners' perceived relationship intimacy levels | within 30 weeks post treatment
  Categorized from the corresponding intimacy scores in the manner of loss of intimacy (0-48), stable relationships (49-71) and improvement (72-120).

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States